CLINICAL TRIAL: NCT02322788
Title: A Randomised, Double-blind, Double-dummy, Multi-site, Phase III, Single Dose, 4-way Cross-over Pharmacodynamic Study Evaluating the Efficacy of Bricanyl Turbuhaler M3 Compared to Bricanyl Turbuhaler M2 by Studying the Protective Effect on Methacholine Induced Bronchoconstriction in Patients With Stable, Mild to Moderate Asthma
Brief Title: Comparing the Efficacy of Bricanyl M2 and Bricanyl M3 at 0.5 and 1.5 mg Dose Levels, to Allow for a Switch From Bricanyl Turbuhaler M2 to Bricanyl Turbuhaler M3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D4711C00001
Record Dates: First submitted 2014-11-26; First posted 2014-12-23 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Inhalation, Pharmacodynamic, Patients,
MeSH Terms: conditions — Asthma; Respiratory Aspiration | interventions — Terbutaline; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bricanyl Turbuhaler M2, Active (Active Comparator): Terbutaline sulphate powder for inhalation, 0.5 mg terbutaline per inhalation
  Interventions: Drug: Terbutaline sulphate
- Bricanyl Turbuhaler M3, Active (Active Comparator): Terbutaline sulphate powder for inhalation, 0.4 mg terbutaline per inhalation
  Interventions: Drug: Terbutaline sulphate
- Turbuhaler M2, Placebo (Placebo Comparator): Placebo powder for inhalation
  Interventions: Drug: Placebo for terbutaline sulphate
- Turbuhaler M3, Placebo (Placebo Comparator): Placebo powder for inhalation
  Interventions: Drug: Placebo for terbutaline sulphate

INTERVENTIONS:
Drug: Terbutaline sulphate — Bricanyl Turbuhaler M2
  Other Names: Terbutaline sulphate powder for inhalation, 0.5 mg (metered dose) terbutaline per inhalation
  Arms: Bricanyl Turbuhaler M2, Active
Drug: Terbutaline sulphate — Bricanyl Turbuhaler M3
  Other Names: Terbutaline sulphate powder for inhalation, 0.4 mg (delivered dose) terbutaline per inhalation
  Arms: Bricanyl Turbuhaler M3, Active
Drug: Placebo for terbutaline sulphate — Placebo Turbuhaler M2
  Other Names: Placebo powder for inhalation
  Arms: Turbuhaler M2, Placebo
Drug: Placebo for terbutaline sulphate — Placebo Turbuhaler M3
  Other Names: Placebo powder for inhalation
  Arms: Turbuhaler M3, Placebo

SUMMARY:
A randomised, double-blind, double-dummy, multi-site, phase III, single dose, 4-way cross-over pharmacodynamic study evaluating the efficacy of Bricanyl Turbuhaler M3 compared to Bricanyl Turbuhaler M2 by studying the protective effect on methacholine induced bronchoconstriction in patients with stable, mild to moderate asthma

DETAILED DESCRIPTION:
The study will include female and male patients, between 18 and 65 years old, with stable, mild to moderate asthma who are on short acting β2-agonist (SABA) alone, on low dose inhaled corticosteroid (ICS) (200-400 µg budesonide or corresponding) or on a combination of low dose ICS and long acting β2-agonists (LABA). Approximately 60 patients will be randomised in order to have 49 completed.

The primary objective is to demonstrate therapeutic equivalence between Bricanyl Turbuhaler M3 and Bricanyl Turbuhaler M2 using bronchoprotective effect. Outcome measure: PC20 (Methacholine provocative concentration causing a 20% drop in FEV1). The safety objective is to compare safety of Bricanyl Turbuhaler M2 and Bricanyl Turbuhaler M3. Outcome measure Adverse Events/Serious.

Study period Q1 2015 - Q1 2016.

ELIGIBILITY:
Inclusion Criteria: - Female and male aged 18 and 65 years.

* At least 6 months of documented clinical diagnosis of asthma as defined by GINA 2012 or American Thoracic Society (Expert Panel Report 3 2007) prior to visit 1
* Stable asthmatics on SABA alone, on low dose ICS (200-400 µg budesonide corresponding) or on fixed combination of low ICS/LABA
* At the enrolment visit 1a, the visit baseline FEV1 must be ≥80 % of that predicted normal (NHANES III). For LABA patients the visit baseline FEV1 must be ≥80 % of that predicted normal (NHANES III) at both visit 1a and visit 1b. If not, the patient will be withdrawn from the study
* At the enrolment visits 1a or 1b (LABA patients only) and at the end of run-in period, visit 2, eligible patients should demonstrate an airway responsiveness to methacholine PC20 <8 mg/mL. If not, the patient will be withdrawn from the study
* Capable of using Turbuhaler inhalation device as judged by investigator. Exclusion Criteria: Diagnosed with COPD or history of cystic fibrosis, bronchiectasis or other respiratory diseases
* Pregnancy, breast-feeding, lactation, or planned pregnancy during the study. Fertile women not using acceptable contraceptive measures
* Conditions which could alter airway reactivity to methacholine (e.g. pneumonia, upper respiratory tract infection, viral bronchitis and/or sinobronchitis) within past six weeks
* Exacerbation due to asthma or change in asthma medication during the last 3 months prior to enrolment
* Night time awakenings due to asthma symptoms on 2 consecutive nights during the last 4 weeks prior to enrolment
* Smokers 6 months prior to the study start or with a history of smoking of more than 10 pack years (e.g. 20 cigarettes/day for at least 10 years, or 10 cigarettes/day for at least 20 years, or equal).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Göran Eckerwall, MD, Study Director — AstraZeneca Mölndal, Sweden; Leif Bjermer, MD, Professor, Principal Investigator — Skånes University hospital, Lund
Locations (4):
- Canada (2):
  - Research Site, Hamilton, Ontario
  - Research Site, Québec, Quebec
- Research Site, Groningen, Netherlands
- Research Site, Lund, Sweden

REFERENCES:
- [Derived] Bjermer L, Gauvreau GM, Postma DS, O'Byrne PM, van den Berge M, Boulet LP, Beckman O, Persson T, Roman J, Carlholm M, Schutzer KM, Eckerwall G. Methacholine challenge tests to demonstrate therapeutic equivalence of terbutaline sulfate via different Turbuhaler(R) devices in patients with mild to moderate asthma: Appraisal of a four-way crossover design. Pulm Pharmacol Ther. 2017 Jun;44:1-6. doi: 10.1016/j.pupt.2017.02.004. Epub 2017 Feb 20. PMID 28232118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with stable, mild to moderate asthma were enrolled. The first subject entered study on March 10, 2015 and the last subject completed study on November 5, 2015. Subjects were recuited from Site 1001 and 1002 in Canada, Site 7201 in Sweden, and Site 5001 in Netherlands.
Pre-assignment Details: Of the 95 patients enrolled 34 were screen failures mainly due to not fulfilling specific randomization criteria on stability in asthma or sensitivity to methacholine challenge; 1 was withdrawal by subject; 72 entered run in period. A total of 60 patients were randomized to the 4 single-dose treatments with terbutaline in a crossover design.
Groups:
- M2 0.5 mg: 0.5 mg terbutaline sulphate administered via Turbuhaler M2
- M2 1.5 mg: 1.5 mg terbutaline sulphate administered via Turbuhaler M2
- M3 0.5 mg: 0.5 mg terbutaline sulphate administered via Turbuhaler M3
- M3 1.5 mg: 1.5 mg terbutaline sulphate administered via Turbuhaler M3
Period: Visit 3
Arm/Group | M2 0.5 mg | M2 1.5 mg | M3 0.5 mg | M3 1.5 mg
Started | 15 | 15 | 14 | 16
Completed | 15 | 15 | 14 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Visit 4
Arm/Group | M2 0.5 mg | M2 1.5 mg | M3 0.5 mg | M3 1.5 mg
Started | 15 | 14 | 16 | 15
Completed | 15 | 14 | 16 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Visit 5
Arm/Group | M2 0.5 mg | M2 1.5 mg | M3 0.5 mg | M3 1.5 mg
Started | 16 | 15 | 15 | 14
Completed | 16 | 15 | 15 | 14
Not Completed | 0 | 0 | 0 | 0
Period: Visit 6
Arm/Group | M2 0.5 mg | M2 1.5 mg | M3 0.5 mg | M3 1.5 mg
Started | 14 | 16 | 15 | 15
Completed | 14 | 16 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Overall: Total number of participants in the Full analysis set
Arm/Group | Overall
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.1 (12.19)
Gender [Count of Participants; unit: Participants]
  Female | 40
  Male | 20
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 57
  Black or African American | 1
  Asian | 2

OUTCOME MEASURES:

1. Primary Outcome: Provocative Concentration of Methacholine Which Produces a 20% Fall in FEV1 (PC20)
Time Frame: 4 cross-over treatments (<1 day each) with 2-10 days between treatment washout periods
Population: Efficacy analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/mL
Arm/Group | M3 1.5 mg | M3 0.5 mg | M2 1.5 mg | M2 0.5 mg
Number analyzed (Participants) | 60 | 60 | 60 | 60
mg/mL | 17.70 [12.51 to 25.05] | 9.88 [6.98 to 13.99] | 20.10 [14.20 to 28.45] | 10.78 [7.61 to 15.25]
Statistical Analysis 1: Comparison: M2 1.5 mg vs M2 0.5 mg; A linear mixed effect model based on restricted maximum likelihood analysis is used to estimate the treatment effect. PC20 in natural log scale is the response variable, treatment and period are the fixed effects, and patient within sequence is a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Estimated mean ratio = 1.87, 95% CI 2-sided [1.52 to 2.29]
Statistical Analysis 2: Comparison: M3 1.5 mg vs M3 0.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Estimated mean ratio = 1.79, 95% CI 2-sided [1.46 to 2.20]
Statistical Analysis 3: Comparison: M3 0.5 mg vs M2 0.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The details of the sample size calculation is document at Section 8.2 the study protocol; Mixed Models Analysis; Estimated mean ratio = 0.92, 95% CI 2-sided [0.75 to 1.13]
Statistical Analysis 4: Comparison: M3 1.5 mg vs M2 1.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The details of the sample size calculation is document at Section 8.2 the study protocol; Mixed Models Analysis; Estimated mean ratio = 0.88, 95% CI 2-sided [0.72 to 1.08]

ADVERSE EVENTS:
Time Frame: During randomized treatment period from Visit 3 to Visit 6
Arm/Group | M2 0.5 mg | M2 1.5 mg | M3 0.5 mg | M3 1.5 mg
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 12/60 | 10/60 | 7/60 | 13/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M2 0.5 mg (N=60) | M2 1.5 mg (N=60) | M3 0.5 mg (N=60) | M3 1.5 mg (N=60)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 6 (6) | 6 (6) | 5 (5) | 7 (7)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1) | 5 (5)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days